CLINICAL TRIAL: NCT04448496
Title: Prospective Trial of Dexamethasone implAnt for Treatment Naïve diabeTic Macular Edema: The Multicenter DANTE Study
Brief Title: Prospective Trial of Dexamethasone implAnt for Treatment Naïve diabeTic Macular Edema
Acronym: DANTE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yeungnam University College of Medicine (Other)
Responsible Party: Principal Investigator, Min Sagong, Professor, Yeungnam University College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YUMC 2020-05-086
Record Dates: First submitted 2020-05-25; First posted 2020-06-26 (Actual); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy | interventions — Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arms (Experimental): Diabetic macular edema Dexamethasone 0.7mg is injected into the vitreous cavity. Center-involved macular edema secondary to diabetic retinopathy for no longer than 3 months (at the screening visit it should be ensured that the subjects will comply with the criterion of ≤ 3 months since onset of macular edema at their scheduled baseline visit)
  Interventions: Drug: Dexamethasone implant

INTERVENTIONS:
Drug: Dexamethasone implant — Dexamethasone 0.7mg is injected into the vitreous cavity through the pars plana using applicator for diabetic macular edema.
  Other Names: Ozurdex

SUMMARY:
The purpose of the investigator's study is to evaluate the efﬁcacy and safety proﬁle of the pro re nata (PRN) regimen to 12 months by using intravitreal dexamethasone implant in eyes with treatment-naive diabetic macular edema patients.

DETAILED DESCRIPTION:
Pathogenesis of diabetic macular edema (DME) involves inflammation, angiogenesis, and oxidative stress processes provoked mainly by cytokines such as interleukin (IL)-6, 8, and monocyte chemotactic protein, and vascular endothelial growth factor (VEGF). Vision loss associated with diabetic retinopathy is most commonly caused by DME, which affects approximately 7% of all diabetic patients. Several therapeutic options are available for treating DME. Evidence for the use of these therapies is accumulating; however, the optical treatment choice remains unclear. In recent years, using intravitreal anti-VEGF agents to treat DME has been shown to be beneficial. Anti-VEGF injections are generally considered suitable first-line therapy for center-involved DME and are effective in improving visual acuity (VA), with 10% to 40% of patients achieving significant improvement in best-corrected visual acuity (BCVA) after 1 year of treatment.

The management of DME is complex, and often multiple treatment approaches are needed. Although anti-VEGF agents were effective for the treatment of DME, there is a proportion of patients who do not achieve optimal response to these agents, presenting refractory or persistent DME. Intravitreal administration of steroids for the treatment of DME has also been studied for many years due to their well-known, widespread, anti-inflammatory effects. Dexamethasone implant is a slow-release dexamethasone delivery system developed for intravitreal administration that has recently been introduced as a therapeutic option in DME.

ELIGIBILITY:
Inclusion Criteria:

1. Male and females 18 years of age or older
2. Written informed consent has been obtained
3. Diabetic macular edema with a central macular thickness (CMT) ≥ 300um measured by spectral domain optical coherence tomography.
4. Treatment-naïve subjects for diabetic macular edema.
5. Documented BCVA of ETDRS letter score of 23 to 73 letters (Snellen equivalent of 20/320 to 20/40) in the study eye.

Exclusion Criteria:

1. Previous panretinal photocoagulation (PRP) or macular laser photocoagulation in the study eye
2. Any prior or concomitant ocular treatment (e.g. anti-VEGF therapy, corticosteroids) in the study eye for diabetic macular edema
3. Prior systemic anti-VEGF or corticosteroid therapy, investigational or approved, within the last 3 months before the first dose in the study
4. Previous use of intraocular corticosteroids in the study eye at any time or use of periocular corticosteroids in the study eye within 12 months prior to Day 1
5. Elevated intraocular pressure or a history of steroid-induced ocular hypertension
6. The presence of other retinopathies, maculopathies, visually signiﬁcant cataract, vitreomacular traction, peripheral ischemia, history of pars plana vitrectomy
7. Any active intraocular, extraocular, and periocular inflammation or infection in either eye within 4 weeks of screening
8. Any history of allergy to povidone iodine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2020-06-22 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean change of best corrected visual acuity | From baseline to month 6
  The mean change of best corrected visual acuity from baseline to Month 6 in early treatment diabetic retinopathy (ETDRS) letter score by using Logarithm of the Minimum Angle of Resolution (LogMAR) chart

SECONDARY OUTCOMES:
Mean change of best corrected visual acuity | From baseline to month 12
  The change in mean best corrected visual acuity at baseline as measured by the early treatment diabetic retinopathy letter score by using Logarithm of the Minimum Angle of Resolution (LogMAR) chart
Mean change in central macular thickness | From baseline to month 6 and 12
  The mean change in central macular thickness (um) by using optical coherence tomography
Mean number of injections | From baseline to month 12
  The mean number of injections
Mean treatment interval between injections | From baseline to month 12
  The mean treatment interval (weeks) between injections
Proportion (%) of subjects who gain ≥ 15 letters in best corrected visual acuity | Compared with baseline at month 6 and 12
  The proportion (%) of subjects who gain ≥ 15 letters in best corrected visual acuity on the early treatment diabetic retinopathy chart
Changes of total area (mm^2)of nonperfusion within the ETDRS grid using fluorescein angiography and optical coherence tomography angiography | From baseline to month 12
  Changes of total area (mm^2) of nonperfusion within the ETDRS grid using fluorescein angiography and optical coherence tomography angiography

CONTACTS AND LOCATIONS:
Overall Officials: Min Sagong, MD,PhD, Principal Investigator — Yeungnam University Hospital
Locations (7):
- South Korea (7):
  - Dong-A University Hospital, Busan
  - Maryknoll Medical Center, Busan
  - Gyeongsang National University Changwon Hospital, Changwon
  - Yeungnam university hospital, Daegu
  - Kyungpook National University Hospital, Daegu
  - Chungnam National University Hospital, Daejeon
  - Chonnam National University Hospital, Gwangju